CLINICAL TRIAL: NCT07023679
Title: The Effect of Targeted Stellate Ganglion Morphine Infiltration on Reperfusion Injury in STEMI Patients After Primary PCI: A Multi-Center Randomized Controlled Trial
Brief Title: Stellate Ganglion Morphine Infiltration on Myocardial I/R Injury
Acronym: tSGM-AMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Ye Zhang, Senior doctor, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YX2025-097
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Acute Myocardial Infarction; Stellate Ganglion; Percutaneous Coronary Intervention; Ischemia/reperfusion injury; Morphine
MeSH Terms: conditions — Reperfusion Injury | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine group (Experimental): Patients in the morphine group will receive a single injection of morphine (10 mg, 10 ml) around the left stellate ganglion under ultrasound guidance before coronary artery recanalization.
  Interventions: Drug: Morphine
- Saline group (Placebo Comparator): Patients in the placebo group will receive a single injection of 0.9% saline (10 ml) around the left stellate ganglion under ultrasound guidance before coronary artery recanalization.
  Interventions: Drug: saline placebo

INTERVENTIONS:
Drug: Morphine — Morphine (10 mg, 10 ml) is injected around the stellate ganglion using ultrasound guidance prior to coronary artery recanalization
  Arms: Morphine group
Drug: saline placebo — Saline (10 ml) is injected around the stellate ganglion using ultrasound guidance prior to coronary artery recanalization
  Arms: Saline group

SUMMARY:
The goal of this clinical trial is to investigate whether morphine modulates the functions of the stellate ganglion to reduce myocardial ischemia/reperfusion (I/R) injury in AMI patients. It will also assess the safety of injecting morphine around the stellate ganglion via ultrasound guidance. The main questions it aims to answer are:

1. Does morphine regulate stellate ganglion function to reduce myocardial I/R injury in AMI patients and improve one year outcome in AMI patients? 3. What medical problems do participants experience when receiving injected morphine around the stellate ganglion? Researchers will compare morphine to a placebo saline (as a control group) to determine whether stellate ganglion infiltration with morphine effectively treats patients with AMI following primary PCI.

Participants will:

* Receive a single injection of morphine or saline around the stellate ganglion.
* Evaluate the myocardial injury during their duration of hospital stay.
* Record their symptoms and any major adverse cardiovascular and cerebrovascular events within one year post-surgery.

DETAILED DESCRIPTION:
Acute ST-segment elevation myocardial infarction (STEMI) patients (aged ≥18 years) planned for percutaneous coronary intervention (PCI) will be eligible for this study. Patients with severe complications of myocardial infarction, such as uncontrollable acute left heart failure or pulmonary edema, severe cardiogenic shock after cardiopulmonary resuscitation, severe mechanical complications including ventricular septal defect, papillary muscle rupture, and rupture of the left ventricular free wall; with old myocardial infarction, or cardiomyopathy, or malignant arrhythmias controlled by antiarrhythmic drugs; with coagulation disorders due to systemic diseases and those who are currently using anticoagulants and are not suitable for injection; with allergy to opioids or with a history of opioid addiction and those participating in other clinical studies; with pregnant or breastfeeding women; with severe organ dysfunction or failure, such as liver failure, renal failure, and respiratory failure; with severe infections; with severe mental illness that cannot cooperate and those taking antipsychotic drugs or considered unsuitable for this study by the researchers will be excluded. Subjects will be randomly assigned to one of two groups: the placebo group and the morphine group. Patients in the morphine group will receive a single injection of morphine (10 mg, 10 ml) around the left stellate ganglion under ultrasound guidance before coronary artery recanalization. Moreover, the placebo group will receive a 10 ml 0.9% saline infiltration around the stellate ganglion. The incidence of major adverse cardiovascular and cerebrovascular events (MACCE) will be recorded within one year post-surgery as the primary outcome. The secondary outcomes include plasma hs-cTnI levels, evaluation of no-reflow phenomenon, major STEMI-related complications within 30 days post-surgery, rehospitalization rate due to cardiovascular adverse events, individual events of MACCE at one year post-surgery or 30 days post-surgery, All-cause mortality, and postoperative hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years, Male or Female.
* Acute ST-segment elevation myocardial infarction (STEMI) patients planned for percutaneous coronary intervention (PCI). Acute STEMI is defined as: electrocardiogram shows ST-segment elevation ≥0.2 mV in two or more adjacent leads, or new left bundle branch block (LBBW).
* Within 24 hours of the onset of infarct-related chest pain.
* Obtaining informed consent from the patient and their family.

Exclusion Criteria:

* Patients with severe complications of myocardial infarction, such as uncontrollable acute left heart failure and pulmonary edema, severe cardiogenic shock after cardiopulmonary resuscitation, severe mechanical complications including ventricular septal defect, papillary muscle rupture, and rupture of the left ventricular free wall;
* Patients with old myocardial infarction, or cardiomyopathy, or malignant arrhythmias controlled by antiarrhythmic drugs;
* Patients with coagulation disorders due to systemic diseases and those who are currently using anticoagulants and are not suitable for injection;
* Patients allergic to opioids or with a history of opioid addiction and those participating in other clinical studies;
* Pregnant or breastfeeding women;
* Patients with severe organ dysfunction or failure, such as liver failure, renal failure, and respiratory failure;
* Patients with severe infections;
* Patients with severe mental illness that cannot cooperate and those taking antipsychotic drugs;
* Other patients considered unsuitable for this study by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2588 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2029-06-20 (Estimated); Study Completion 2029-06-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of major adverse cardiovascular and cerebrovascular events (MACCE) | within one year post-surgery
  The incidence of major adverse cardiovascular and cerebrovascular events (MACCE), defined as cardiac death, heart failure rehospitalization, recurrent myocardial infarction, coronary revascularization, and stroke, will be recorded within one year post-surgery.

SECONDARY OUTCOMES:
Postoperative plasma hs-cTnI levels | at 24 hours post-surgery
  The levels of plasma hs-cTnI will be recorded at 24 hours post-surgery.
Evaluation of no-reflow phenomenon | perioperative
  The S-T segment deviation is measured as the height difference (in millimeters) between the J point and the baseline ( the PR segment) at 2 hours, 24 hours, and either discharge or 7 days post-surgery.
Major STEMI-related complications within 30 days post-surgery | within 30 days post-surgery
  The major STEMI-related complications, including cardiogenic shock, acute left heart failure, mechanical complications, malignant arrhythmias, will be recorded within 30 days post-surgery.
Rehospitalization rate due to cardiovascular adverse events | within one year post-surgery
  The rehospitalization rate due to cardiovascular adverse events will be recorded within one year post-surgery.
All-cause mortality | within one year post-surgery
  All-cause mortality will be recorded within one year post-surgery.
Individual events of MACCE at one year post-surgery or 30 days post-surgery | within one year post-surgery or 30 days post-surgery
  The individual event of MACCE will be recorded at one year post-surgery or 30 days post-surgery
Postoperative hospital stay | Perioperative
  The length of the postoperative hospital stay will be determined by the duration from the completion of surgery to discharge.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei